CLINICAL TRIAL: NCT05333133
Title: High Calorie Formula Intervention on Weight, Length, Total Lymphocyte Count, TNF-α and IGF-1 in Growth Faltering Children
Brief Title: High Calorie Formula Intervention on Weight, Length Increment, Total Lymphocyte Counts, TNF-alpha and IGF-1 in Failure to Thrive Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Airlangga (Other)
Collaborators: Danone Institute International (Other)
Responsible Party: Principal Investigator, Andy Darma, MD, Principal Investigator on Gastroenterology, Universitas Airlangga
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IGF-1 in failure to thrive
Record Dates: First submitted 2022-03-25; First posted 2022-04-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Failure to Thrive; Infection, Bacterial; Growth Faltering
MeSH Terms: conditions — Failure to Thrive; Bacterial Infections | interventions — Food, Formulated

STUDY DESIGN:
Intervention Model Description: Pre-, post- intervention study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High calorie formula on IGF-1, TNF-alpha and total lymphocyte counts (Experimental): Interventional study with pre-, post design after the subjects are diagnosed with TB and UTI, they will receive 400 ml (equal with 400 kcal) of high calorie formula per day, prescribed by the researcher (a pediatrician) for 90 days consumption. Body weight and body height will be monitored by the researcher group every 30 days to record the tolerance, acceptance and complaints (and the side effects) the blood will be withdraw at day 0 (before intervention) and day 90 (after intervention) to investigate the IGF-1, TNF-alpha and total lymphocyte counts
  Interventions: Dietary Supplement: high calorie formula (oral nutritional supplement/ONS)

INTERVENTIONS:
Dietary Supplement: high calorie formula (oral nutritional supplement/ONS) — every subject is given 400 ml (equal with 400 kcal) high calorie formula for 90 days. before (day 0) and after (day 91) the intervention was enrolled, blood samples was taken to investigate IGF-1 and total lymphocyte counts.
  The body weight and body height will be measured at day-0, day-14, day-30, day 60 and 90.
  Other Names: formula for special medical purposes

SUMMARY:
High calorie formula (Oral Nutrition Supplement/ONS) are products used for oral nutrition support with the aim to increase the nutritional intake. they are a nutrition treatment option children with limited intake. ONS are typically used in addition to a normal diet, when diet alone is insufficient to meet daily nutritional requirement due to infection or others. ONS should be treated like medication, ensure they are labelled with the patient's name and provided at the prescribed time.

It is well established that nutritional deficiency or inadequate can impair immune function. Growing evidence suggest that for certain conditions, the nutrient needs will be increased, so it is needed to provide the nutrient intake above currently recommended levels, in order to help optimizing the immune function, including improving the defense function and thus resistance to infection while maintaining tolerance.

Purposes:

1. to analyze the effect of high calorie formula on IGF-1 levels in children with failure to thrive
2. to analyze the effect of high calorie formula on total lymphocyte counts with failure to thrive
3. to analyze the effect of high calorie formula on TNF-alpha levels in children with failure to thrive

Hypothesis:

1. there is significant increment of IGF-1 levels before and after the intervention
2. there is significant difference of total lymphocyte counts before and after the intervention
3. there is significant difference of TNF-alpha levels before and after the intervention

DETAILED DESCRIPTION:
Interventional study with pre-, post-test design. After the subject were diagnosed with infection (tuberculosis/TB or urinary tract infection/ UTI, the diagnosed will be determined by a pediatrician/the researcher based on clinical examination and laboratory findings), they will receive 400 kcal/day (96 g/day divided 4 times consumption) of high calorie formula prescribed by the researcher (A pediatrician) for 90 days consumption (8640 g). the subject will monitored every 30 days for acceptance, tolerance, weight increment, length increment evaluation until the end of study (90 day intervention).

The blood will be withdrawn at day 0 (before invention) and day 90 (after intervention) to measure the levels of TNF-alpha, IGF-1 and total lymphocyte count. Total lymphocyte count (TLC) was measured based on the complete blood report (white blood cells x 1000 x % lymphocyte). The high calorie formula is given as much as 400 kcal/day for 90 days after the subject were diagnosed with tuberculosis (TB) or urinary tract infection (UTI), determine as day 1. Before the intervention (day 0) and after the intervention (day 90), the subjects were taken the blood by laboratory employee of the private hospital in Surabaya, Indonesia.

The statistical analysis including test of normality and homogeneity test, followed by paired sample T-test or Wilcoxon, depend on the normality and homogeneity test.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 years - 5 years, are diagnosed tuberculosis (TB) and urinary tract infection (UTI)

Exclusion Criteria:

* Congenital Disease
* Congenital Heart Disease
* Edema
* Organomegaly
* Tumor
* Cerebral palsy and genetic syndromes
* Hormonal abnormality/disorders

Drop out criteria:

* Lost contact

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
The effectiveness of high calorie formula on the subjects | 90 days
  Change on body weight. The data will be presented as mean +/- SD (standard deviation). The body weight will be measure with baby Scale Seca 354 (in grams) for subjects <24 months age, and using Seca electronic flat scale 813 (in grams) for subjects >24 months age
The effectiveness of high calorie formula on the subjects | 90 days
  Change on body height/length. The data will be presented as mean +/- SD (standard deviation). The body height/length will be measure with infantometer Seca 416 (in cm) for subject <24 months age, and using stadiometer Seca 213 (in cm) for subjects >24 months age
The effectiveness of high calorie formula on the subjects | day 0 pre intervention, day 91 post intervention
  Change on IGF-1 levels (in ng/ml) will be presented as mean +/- SD (standard deviation). IGF-1 levels will be measured using Human IGF-1 Elisa kit 96 T (BT LAB),
The effectiveness of high calorie formula on the subjects | 90 days
  The change on total lymphocyte count (TLC) before and after intervention, the data will be presented as mean +/- SD (standard deviation). TLC will measure based on complete blood count (CBC), with formula WBC x 1000 x % lymhocyte, express as a decimal.

SECONDARY OUTCOMES:
The effectiveness of high calorie formula on the subjects | 90 days
  Change on TNF-alpha levels (in ng/ml) will be presented as as mean +/- SD (standard deviation). TNF-alpha will measure using Human TNF-alpha Elisa kit 96 T (BT LAB).

CONTACTS AND LOCATIONS:
Locations (1):
- Husada Utama Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No